CLINICAL TRIAL: NCT06036888
Title: DEFILE-QoL5 - Evaluation de la Prise en Charge Chirurgicale à 5 Ans du Syndrome du défilé Thoraco-brachial
Brief Title: DEFILE-QoL5 - Evaluation of the Long-term Surgical Management of the Thoraco-brachial Displacement Syndrome
Acronym: DEFILE-QoL5
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2023-A00126-39
Record Dates: First submitted 2023-08-29; First posted 2023-09-14 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Thoracic Outlet Syndrome
MeSH Terms: conditions — Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- thoracobrachial outlet syndrome: Patient :
  * adult
  * with thoraco-brachial outlet syndrome
  * who has participated to DEFILE-QoL study in 2016
  * who accept to participate and is able to complete questionaries
  Interventions: Other: questionaries completion

INTERVENTIONS:
Other: questionaries completion — Answer to the DASH and SF-12 questionaries, for an estimated duration of 15 minutes.

SUMMARY:
The study concerns patients hospitalized in vascular and thoracic surgery in 2016 at the University Hospital of Angers for the management of a thoraco-brachial outlet syndrome. It includes all vascular and neurological manifestations related to intermittent or permanent compression of the vasculo-nervous bundle of the upper limb. Before and after the operation, these patients had agreed to complete the quality of life questionnaires, the Disabilities of the Arm, Shoulder and Hand questionary (DASH) and the Short-Form 12 (SF-12). The objective of the present study is to evaluate the long-term quality of life, using the questionnaires mentioned above, completed by 54 patients treated surgically for thoraco-brachial outlet syndrome and who participated in the DEFILE-QoL study in 2016.

DETAILED DESCRIPTION:
All patients included in the DEFILE-QoL study (in 2016) receive an information letter. Without opposition from them after 4 weeks, they are contacted by telephone. The telephone interview begins with an explanation of the study and a time to answer any questions from the patient.

If they agree to participate, they answer the DASH and the SF-12 questionnaires, for an estimated duration of 15 minutes. Following the telephone interview, the patient's participation in the study was terminated.

The date of the information and the patient's non-objection are documented in the patient's source file.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* having participated in the initial study : "DEFILE-QoL"

Exclusion Criteria:

* opposing participation in the research
* unable to answer questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for thoraco-brachial outlet syndrome and treated surgically in the department of university Angers hospital in 2016
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Quality of life scores | at least 5 years after surgery
  Assess the quality of life, using standardized questionnaires, of patients treated surgically for thoraco-brachial outlet syndrome

SECONDARY OUTCOMES:
Factors associated with poor long-term clinical outcome | at least 5 years after surgery
  Identify factors associated with poor long-term clinical outcome (DEFILE-QoL in 2016) : clinical presentation of Syndrome, its severity, the imaging examinations performed and the various scores collected

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Jaglin-Grimonprez, Study Director — University hospital of Angers
Locations (1):
- Myriam AMMI, Angers, Maine Et Loire, France